CLINICAL TRIAL: NCT06875492
Title: Retrospective Cohort Study on the Impact of PDL Treatment History on the Efficacy of HMME-PDT in Treating PWS Children
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Other Study IDs: 2024218
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Port-Wine Stain
Keywords: Pulse dye laser; Hemoporfin-PDT
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1 (No PDL): Cohort 1 (No PDL) comprised patients without a history of PDL treatment
  Interventions: Combination Product: HMME-PDT
- Cohort 2 (Prior PDL): Cohort 2 (Prior PDL) consisted of patients with a history of PDL treatment
  Interventions: Combination Product: HMME-PDT; Device: PDL

INTERVENTIONS:
Combination Product: HMME-PDT — Twice HMME-PDT, and the treatment interval is 2 to 3 months.
Device: PDL — Prior PDL treatment history.
  Groups: Cohort 2 (Prior PDL)

SUMMARY:
This retrospective study investigated the influence of prior pulse dye laser (PDL) treatment on the effectiveness of Hemoporfin-PDT in young children aged 1-3 years with PWS.

The study population included patients without a history of PDL treatment and patients with a history of PDL treatment.

DETAILED DESCRIPTION:
Background Hemoporfin-mediated photodynamic therapy (Hemoporfin-PDT) is considered a safe and effective treatment for port-wine stains (PWS). This study aims to investigate the influence of prior pulse dye laser (PDL) treatments history on the effectiveness of Hemoporfin-PDT in young children aged 1-3 years with PWS.

Methods Data was gathered for individuals with PWS aged 1-3 years who received two or more Hemoporfin-PDT treatments. The study population was stratified into two groups: Cohort 1 (No PDL) comprised patients without a history of PDL treatment, while Cohort 2 (Prior PDL) consisted of patients with a history of PDL treatment. An analysis was conducted to investigate the relationship between treatment efficacy and variables including gender, age, location, and type of PWS.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with PWS (Port Wine Stain) who were between 1 and 3 years old at the time of their first HMME-PDT treatment.

  * Patients who, after evaluation by a clinician, are deemed eligible for HMME-PDT treatment and whose guardians have signed an informed consent form.

    * Patients who have undergone two or more HMME-PDT treatments.

      ④ Patients with complete basic information and treatment-related information.

Exclusion Criteria:

* Exclusion of patients with syndromes associated with PWS.

  * Exclusion of patients with a history of treatments for PWS other than PDL treatment.

    * Patients with other vascular malformations. ④ Exclusion of patients who have received any other PWS treatment within 2 months prior to HMME-PDT treatment.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This cohort study is a retrospective, single-center study based on a database established by the photodynamic therapy team at the Second Affiliated Hospital of Xi'an Jiaotong University.We defined "young children" as children aged 1 to 3 years. This research encompassed young children who had undergone two or more sessions of Hemoporfin-PDT. Data on gender, age, medical history, type of PWS, lesion location, and post-treatment efficacy were collected following two rounds of Hemoporfin-PDT.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The rate of lesions regression | The efficacy evaluation will be conducted 3 months after the completion of the 2nd HMME-PDT treatment.
  Two independent blinded assessors assessed treatment efficacy by comparing before and after treatment photos of patients receiving Hemoporfin-PDT for reducing redness. The final outcome was determined as the average of these two assessments. Efficacy was assessed using standard quartiles: Excellent (76-100 %); Good (51-75 %); Fair (26-50 %); Poor (0-25 %).

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No